CLINICAL TRIAL: NCT02616003
Title: A Novel Preoperative Conditioning Therapy in Giant Obese Patients With the Combination of Liraglutide and a Leucine-Based Amino-Acid Infusion and Caloric Restriction
Brief Title: Preoperative Condition in Giant Obese Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sana Klinikum Offenbach (Other)
Responsible Party: Principal Investigator, Christine Stier, MD, PhD, Sana Klinikum Offenbach
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FF 121/2015
Record Dates: First submitted 2015-11-17; First posted 2015-11-26 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Morbid Obesity; Bariatric Surgery Candidate
Keywords: Morbid Obesity; Giant Obese; Preoperative Procedure; Liraglutide; Leucine
MeSH Terms: conditions — Obesity, Morbid | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Super-super Obese Patients (Other): Multimorbid, super-super obese patients that need preoperative conditioning therapy (intervention 1: Liraglutide, intervention 2: aminosteril hepa 8%, intervention 3: Caloric diet with 1000 kcal) for weight loss surgery to achieve technical operability.
  Interventions: Drug: Liraglutide; Other: Aminosteril hepa 8%; Dietary Supplement: Caloric diet with 1000 kcal

INTERVENTIONS:
Drug: Liraglutide — Initially 1.2 mg Liraglutide as subcutaneous daily injection, boosted to 1.8 mg Liraglutide after 3 days subsequently. 1000 ml infusion of aminosteril hepa 8% from day 1 onwards. Caloric diet with 800 kcal from day 1 onwards till technical operability is achieved (about 21 days)
  Other Names: Victoza
Other: Aminosteril hepa 8% — Initially 1.2 mg Liraglutide as subcutaneous daily injection, boosted to 1.8 mg Liraglutide after 3 days subsequently. 1000 ml infusion of aminosteril hepa 8% from day 1 onwards. Caloric diet with 800 kcal from day 1 onwards till technical operability is achieved (about 21 days)
Dietary Supplement: Caloric diet with 1000 kcal — Initially 1.2 mg Liraglutide as subcutaneous daily injection, boosted to 1.8 mg Liraglutide after 3 days subsequently. 1000 ml infusion of aminosteril hepa 8% from day 1 onwards. Caloric diet with 1000 kcal from day 1 onwards till technical operability is achieved (about 21 days)

SUMMARY:
The frequency of super-super obese who need immediate weight loss surgery is risen continuously. For those patients a prior-to-surgery conditioning therapy is mandatory to gain technical and physical operability. The exclusively well-established preliminary therapy so far was the intragastric balloon, which takes 7 months of treatment time. Due to life-threatening conditions of giant obese patients, who have been admitted to hospital, the investigators were forced to develop a more prompt acting conditioning therapy to bring those individuals in a short run to an improved and "fit-for-surgery" state. In such an impasse the investigators combine Liraglutide with its well-known weight-loss effect with a leucine-based amino acid infusion that is generally used for patients with liver insufficiency, in expectance of an additional weight loss and liver reduction effect.

DETAILED DESCRIPTION:
The investigators will use a commercial available amino acid infusion (Aminosteril hepa 8%, Fresenius Karbi), which is used in clinical application for liver conditioning. It is mainly based on the branched-chained amino acid leucine (13.09 g per 1000 ml). The investigators will combine this with a daily subcutaneous injection of Liraglutide. Liraglutide is a GLP-1 analogue, which achieved meanwhile the FDA approval for weight loss treatment. Initial Liraglutide dosage is 1.2 mg for three days, boosted to 1.8 mg consecutively. Participants receive energy reduced nutrition with 1000 kcal/d.

ELIGIBILITY:
Inclusion Criteria:

* multimorbid, super-super obese patients

Exclusion Criteria:

* renal insufficiency III

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Operability | 21 days
  Operability means that weight loss surgery could be performed after preoperative condition (due to less visceral fat, less liver volume)

SECONDARY OUTCOMES:
Chronic inflammation | 21 days
  Changing in CRP in g/l during intervention
Chronic inflammation II | 21 days
  Changing in white blood cell count /nl during intervention
Liver volume | 21 days
  Changing of liver volume during intervention measured by ultrasound
Liver function | 21 days
  Changing of GOT in U/l, GPT in U/l, GGT in U/l and AP in U/l
Pulmonary function | 21 days
  Changing in FEV1 in lung function testing during intervention
Hg A1c in % | 21 days
Total Protein in g/l | 21 days
Preoperative excess weight loss in % | 21 days
Albumin in g/l | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Weiner, MD, Prof., Study Chair — Sana Klinikum Offenbach
Locations (1):
- Sana Klinikum Offenbach, Offenbach, Hesse, Germany

REFERENCES:
- [Result] Baggio LL, Drucker DJ. Glucagon-like peptide-1 receptors in the brain: controlling food intake and body weight. J Clin Invest. 2014 Oct;124(10):4223-6. doi: 10.1172/JCI78371. Epub 2014 Sep 9. PMID 25202976
- [Result] Alhadeff AL, Baird JP, Swick JC, Hayes MR, Grill HJ. Glucagon-like Peptide-1 receptor signaling in the lateral parabrachial nucleus contributes to the control of food intake and motivation to feed. Neuropsychopharmacology. 2014 Aug;39(9):2233-43. doi: 10.1038/npp.2014.74. Epub 2014 Mar 26. PMID 24681814
- [Result] Pi-Sunyer X, Astrup A, Fujioka K, Greenway F, Halpern A, Krempf M, Lau DC, le Roux CW, Violante Ortiz R, Jensen CB, Wilding JP; SCALE Obesity and Prediabetes NN8022-1839 Study Group. A Randomized, Controlled Trial of 3.0 mg of Liraglutide in Weight Management. N Engl J Med. 2015 Jul 2;373(1):11-22. doi: 10.1056/NEJMoa1411892. PMID 26132939
- [Result] Pedroso JA, Zampieri TT, Donato J Jr. Reviewing the Effects of L-Leucine Supplementation in the Regulation of Food Intake, Energy Balance, and Glucose Homeostasis. Nutrients. 2015 May 22;7(5):3914-37. doi: 10.3390/nu7053914. PMID 26007339
- [Result] Zhang Y, Guo K, LeBlanc RE, Loh D, Schwartz GJ, Yu YH. Increasing dietary leucine intake reduces diet-induced obesity and improves glucose and cholesterol metabolism in mice via multimechanisms. Diabetes. 2007 Jun;56(6):1647-54. doi: 10.2337/db07-0123. Epub 2007 Mar 14. PMID 17360978
- [Result] McAllan L, Cotter PD, Roche HM, Korpela R, Nilaweera KN. Impact of leucine on energy balance. J Physiol Biochem. 2013 Mar;69(1):155-63. doi: 10.1007/s13105-012-0170-2. Epub 2012 Apr 26. PMID 22535285
- [Derived] Stier C, Koschker AC, Kim M, Stier R, Chiappetta S, Stein J. Fast-track rescue weight reduction therapy to achieve rapid technical operability for emergency bariatric surgery in patients with life-threatening inoperable severe obesity - A proof of concept study. Clin Nutr ESPEN. 2022 Aug;50:238-246. doi: 10.1016/j.clnesp.2022.05.009. Epub 2022 May 26. PMID 35871930